CLINICAL TRIAL: NCT07133724
Title: Digital Health for Aging: A Multimodal AI-Based Smart Assessment and Rehabilitation Training System for Lumbar Degeneration
Brief Title: Digital Health for Lumbar Degeneration
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202502072RIND
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Degenerative Lumbar Spine Diseases
Keywords: degenerative lumbar spine disease; real-time detection; artificial Intelligence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-Based Smart Assessment and Rehabilitation Training (Experimental): The multimodal AI-based smart assessment and rehabilitation training system developed in this study will provide patients with lumbar degeneration a convenient and precise home-based rehabilitation solution.
  Interventions: Other: AI-Based Smart Assessment and Rehabilitation Training

INTERVENTIONS:
Other: AI-Based Smart Assessment and Rehabilitation Training — Through the integration of wireless inertial sensors and smartphone imaging, the system can monitor pelvic and lumbar movements in real time, generate a digital twin model, and deliver instant feedback to guide patients in performing correct exercises.

SUMMARY:
This study will integrate wireless wearable sensors, smartphone imaging, and multimodal artificial intelligence (AI) to address the rehabilitation needs of patients with lumbar degeneration. Patients will undergo comprehensive functional assessments, and individualized exercise instruction with real-time feedback will be provided through a smartphone application. The goals of this research are to: (1) develop a multimodal AI-based digital health system combining IMU sensors and smartphone cameras for real-time assessment and interactive rehabilitation training, (2) construct biomechanics- and gait-analysis models to support personalized rehabilitation for patients with lumbar degeneration, and (3) investigate the mechanisms and clinical efficacy of pelvic control exercise training combined with real-time smartphone feedback in improving function and quality of life for aging patients.

DETAILED DESCRIPTION:
The multimodal AI-based smart assessment and rehabilitation training system developed in this study will provide patients with lumbar degeneration a convenient and precise home-based rehabilitation solution. Through the integration of wireless inertial sensors and smartphone imaging, the system can monitor pelvic and lumbar movements in real time, generate a digital twin model, and deliver instant feedback to guide patients in performing correct exercises. This design not only improves patients' self-awareness of posture and movement but also reduces the risk of improper compensatory strategies that often occur in traditional home exercise programs.

The system is particularly suitable for older adults with mobility limitations or those who have difficulties frequently visiting medical institutions. By enabling remote assessment, individualized training, and long-term monitoring, this platform ensures continuity of care and enhances patients' motivation to engage in rehabilitation. The outcomes of this project will establish a tele-rehabilitation system tailored to degenerative lumbar spine disease, support clinicians in delivering precise and effective treatment, and ultimately reduce the healthcare and economic burden on families and society.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 50-80 years to capture the typical characteristics of lumbar degeneration in this age group.
2. No history of low back pain lasting more than one week or severe enough to interrupt work within the past year.
3. Normal lumbar functional mobility.
4. Ability to walk independently for more than 10 meters.

Exclusion Criteria:

1. Presence of systemic joint diseases such as ankylosing spondylitis, rheumatoid arthritis, or multiple sclerosis, which may significantly affect lumbar mobility and gait patterns.
2. Central nervous system disorders (e.g., spinal cord injury, stroke, or Parkinson's disease) that may influence gait and motor control.
3. Vestibular system disorders, to avoid balance abnormalities interfering with gait testing.
4. History of spinal or lower limb surgery, as postoperative changes may affect the accuracy of gait data.
5. Inability to communicate or follow instructions.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional assessment: Walking speed | 6 months
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking speed (unit: m/s).
Functional assessment: Walking distance | 6 months
  Functional assessment is a process that allows for the identification of disability. The data from the functional assessment is used to calculate walking distance (unit: m).
Functional assessment: 5 Times Sit to Stand Test | 6 months
  Functional assessment is a process that allows for the identification of disability. The data from the 5 Times Sit to Stand Test is used to calculate the duration it took to complete the test (unit: s).

SECONDARY OUTCOMES:
Kinematic variables: Joint angles | 6 months
  A motion capture system is used to measure the joint kinematics. The data is used to calculate joint angles (unit: degree).
Kinetic variables | 6 months
  A motion capture system is used to measure the joint kinetics. The data is used to calculate joint moments (unit: Nm)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan